CLINICAL TRIAL: NCT04265677
Title: FamilyLink Family-Centered Rounds Pilot Study
Brief Title: FamilyLink Family-Centered Rounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1524392
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Family Centered Rounds
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine FCR (Experimental): These patients will be eligible to use telemedicine for Family Centered Rounds
  Interventions: Other: Telemedicine FCR
- Control (Placebo Comparator): These patients will not be eligible to use telemedicine for Family Centered Rounds (standard of care)
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Telemedicine FCR — Parents/guardians will be able to join family centered rounds using telemedicine (audio and visual)
  Arms: Telemedicine FCR
Other: Standard of care — Parents/guardians will not be able to join family centered rounds using telemedicine (audio and visual)
  Arms: Control

SUMMARY:
This study will be a pilot test of using FamilyLink software to bring parents of patients in the neonatal intensive care unit (NICU) virtually to the bedside during Family Centered Rounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Blue Team in the NICU aged 0-365 days
* Parents/guardians of patients admitted to the Blue Team in the NICU aged ≥ 18 years
* Medical team members (physicians, nurse practitioners, fellows, residents, medical students, nurses) of patients admitted to the Blue Team in the NICU aged ≥ 18 years

Exclusion Criteria:

* Patients who are not discharged home from the NICU (e.g., transferred to another inpatient unit or another hospital)
* Parents/guardians of patients admitted to the Blue Team in the NICU who do not speak English, as a translator will not reliability be available to participate in rounds when the parent/guardian is not physically present
* Patients who have more than one admission to the Blue Team during our study period will only be included on their first admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
CAHPS Communication with Parent Subscale | Through study completion, approximately 3 months
  19 questions from the Communication with Parent Subscale of the Consumer Assessment of Healthcare Providers and Systems Child Hospital Survey; specifically, we will report the following measures: Communication between you and your child's nurses (composite measure); Communication between you and your child's doctors (composite measure); Communication about your child's medicines (composite measure); Keeping you informed about your child's care (composite measure) Privacy when talking with doctors, nurses, and other providers (single-item measure); Preparing you and your child to leave the hospital (composite measure); Keeping you informed about your child's care in the Emergency Room (single-item measure). Higher scores are better; 0 (minimum) - 100 (maximum)

SECONDARY OUTCOMES:
Rates of adverse events | Up to 6 months
  Rates of adverse events reported by parents, providers, or nurses
Hospital Length of Stay | Through study completion, approximately 3 months
  Hospital length of stay of the patient measured in days
Breastmilk at discharge | Through study completion, approximately 3 months
  If the patient was receiving all, some or no breastmilk

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No